CLINICAL TRIAL: NCT06674629
Title: Effects of an Asymmetrical High Flow Nasal Cannula Interface on End-Expiratory Lung Impedance
Brief Title: Asymmetrical High Flow Nasal Cannula and End-Expiratory Lung Impedance
Acronym: EELI and AHFNC
Status: Completed | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Hospital Británico de Buenos Aires, Argentinian Intensive Care Society
Other Study IDs: #30102024
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: End-Expiratory Lung Impedance; Respiratory Rate; Diaphragm Thickness Fraction; Diaphragm Excursion
Keywords: High Flow Oxygen Therapy; End-Expiratory Lung Impedance; Respiratory rate; Diaphragm Thickness Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteers: Healthy adult volunteers, all above 18 years of age, who provide informed consent.
  Interventions: Device: High flow oxygen therapy

INTERVENTIONS:
Device: High flow oxygen therapy — Application of high flow oxygen therapy through asymmetric cannula at 40 and 60 L/m

SUMMARY:
Objective: The primary aim is to assess end-expiratory lung impedance (EELI) changes during the application of high-flow oxygen therapy using asymmetric nasal cannulae, comparing conditions with the mouth closed and open in healthy volunteers in various positions. The secondary objective includes evaluating respiratory rate, shortening fraction, and diaphragm excursion via ultrasound.

Study Design: This is a prospective observational cohort study conducted in the Critical Care Unit of Sanatorio Parque Rosario from November 5 to December 31, 2024. It will involve 20 healthy adult volunteers without respiratory conditions, with informed consent obtained from all participants. Volunteers with contraindications for electrical impedance tomography (EIT) will be excluded.

Methods: Equipment Used: PulmoVista 500 Dräger (EIT), AIRVO 2 (high-flow oxygen generator), asymmetric nasal cannula (Optiflow OPT 966), Toshiba iStyle ultrasound machine.

Procedures: The study includes EELI measurements in different positions (semi-seated, supine Fowler, prone, and prone Fowler) with various high-flow oxygen settings (40 and 60 L/min). Diaphragm excursion and thickening will be assessed using ultrasound.

Scenarios and Measurements: 17 different testing scenarios will be conducted, with 16 intervals for washout breathing at room air between scenarios. Data on EELI, respiratory rate, and diaphragm measurements will be collected.

DETAILED DESCRIPTION:
Methodology:

Procedures: EELI, respiratory rate, and diaphragm measurements will be taken in various body positions while using high-flow oxygen therapy (HFNC) set at 40 and 60 L/min. Diaphragm excursion and thickening will be evaluated with ultrasound.

Data Collection and Analysis: Volunteers will participate in 17 different testing scenarios, with intervals of 5-minute washout periods breathing room air in a semi-seated position between each measurement. Continuous variables will be expressed as mean ± standard deviation or median and interquartile range. Repeated measures ANOVA will be used for statistical comparisons, with significance set at p < 0.05.

17 Testing Scenarios:

Semi-seated at 45° breathing room air. Semi-seated at 45° with asymmetric HFNC at 40 L/min, mouth closed for 5 minutes.

Semi-seated at 45° with asymmetric HFNC at 40 L/min, mouth open for 5 minutes. Semi-seated at 45° with asymmetric HFNC at 60 L/min, mouth closed for 5 minutes.

Semi-seated at 45° with asymmetric HFNC at 60 L/min, mouth open for 5 minutes. Supine in Fowler position (60°) with asymmetric HFNC at 40 L/min, mouth open for 5 minutes.

Supine in Fowler position (60°) with asymmetric HFNC at 40 L/min, mouth closed for 5 minutes.

Supine in Fowler position (60°) with asymmetric HFNC at 60 L/min, mouth open for 5 minutes.

Supine in Fowler position (60°) with asymmetric HFNC at 60 L/min, mouth closed for 5 minutes.

Prone at 180° with asymmetric HFNC at 40 L/min, mouth open for 5 minutes. Prone at 180° with asymmetric HFNC at 40 L/min, mouth closed for 5 minutes. Prone at 180° with asymmetric HFNC at 60 L/min, mouth open for 5 minutes. Prone at 180° with asymmetric HFNC at 60 L/min, mouth closed for 5 minutes. Prone Fowler position with asymmetric HFNC at 40 L/min, mouth open for 5 minutes.

Prone Fowler position with asymmetric HFNC at 40 L/min, mouth closed for 5 minutes.

Prone Fowler position with asymmetric HFNC at 60 L/min, mouth open for 5 minutes.

Prone Fowler position with asymmetric HFNC at 60 L/min, mouth closed for 5 minutes.

Duration per Participant: Approximately 2 hours and 15 minutes.

Ethical Considerations: All data will be anonymized and kept confidential. Participants' rights to withdraw at any time will be respected, and no personal identifying information will be disclosed.

This comprehensive approach aims to elucidate the physiological impacts of using asymmetric HFOT on end-expiratory lung volume and related respiratory parameters in various positions and conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between 18 and 50 years of age who sign the informed consent form, without respiratory pathology.

Exclusion Criteria:

* contraindication to implement electrical impedance tomography or high flow oxygen therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers healthcare professionals working at Sanatorio Parque in Rosario, aged between 18 and 50 years, who sign the informed consent form and have no history of respiratory pathology (who are non-smokers and do not have a history of any type of respiratory disease).
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
End-Expiratory Lung Impedance | From enrollment to the end of treatment at 2.30hours
  Variation of end-expiratory lung impedance in different positions and with different flows.

SECONDARY OUTCOMES:
Respiratory Rate | From enrollment to the end of treatment at 2.30hours
  Number of respiratory cycles per minute while breathing in a quiet manner at rest.
Diaphragm Thickness Fraction | From enrollment to the end of treatment at 2.30hours
  Diaphragm Thickness Fraction (DTF) is a measure used to assess diaphragm function by comparing the change in diaphragm thickness from end-expiration to end-inspiration expressed as a percentage
Diaphragm excursion | From enrollment to the end of treatment at 2.30hours
  Diaphragm excursion refers to the movement or displacement of the diaphragm during the respiratory cycle, measured from its lowest position at end-expiration to its highest position at end-inspiration. This parameter is assessed using ultrasound and reflects the diaphragm's ability to contract effectively, with greater excursion indicating stronger respiratory muscle function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Británico de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
all IPD on which the results of the publication are based will be in the publication or shared through direct links after consultation with the PI via e-mail
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2025-January 2026

REFERENCES:
- [Background] Slobod D, Spinelli E, Crotti S, Lissoni A, Galazzi A, Grasselli G, Mauri T. Effects of an asymmetrical high flow nasal cannula interface in hypoxemic patients. Crit Care. 2023 Apr 18;27(1):145. doi: 10.1186/s13054-023-04441-6. PMID 37072854
- [Background] Boscolo A, Pettenuzzo T, Zarantonello F, Sella N, Pistollato E, De Cassai A, Congedi S, Paiusco I, Bertoldo G, Crociani S, Toma F, Mormando G, Lorenzoni G, Gregori D, Navalesi P. Asymmetrical high-flow nasal cannula performs similarly to standard interface in patients with acute hypoxemic post-extubation respiratory failure: a pilot study. BMC Pulm Med. 2024 Jan 8;24(1):21. doi: 10.1186/s12890-023-02820-x. PMID 38191347
- [Background] Tatkov S, Rees M, Gulley A, van den Heuij LGT, Nilius G. Asymmetrical nasal high flow ventilation improves clearance of CO2 from the anatomical dead space and increases positive airway pressure. J Appl Physiol (1985). 2023 Feb 1;134(2):365-377. doi: 10.1152/japplphysiol.00692.2022. Epub 2023 Jan 12. PMID 36633864
- [Background] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Background] Parke RL, Eccleston ML, McGuinness SP. The effects of flow on airway pressure during nasal high-flow oxygen therapy. Respir Care. 2011 Aug;56(8):1151-5. doi: 10.4187/respcare.01106. Epub 2011 Apr 15. PMID 21496369
- [Background] Groves N, Tobin A. High flow nasal oxygen generates positive airway pressure in adult volunteers. Aust Crit Care. 2007 Nov;20(4):126-31. doi: 10.1016/j.aucc.2007.08.001. Epub 2007 Oct 10. PMID 17931878
- [Background] Plotnikow GA, Thille AW, Vasquez DN, Pratto RA, Quiroga CM, Andrich ME, Dorado JH, Gomez RS, D'Annunzio PA, Scapellato JL, Intile D. Effects of High-Flow Nasal Cannula on End-Expiratory Lung Impedance in Semi-Seated Healthy Subjects. Respir Care. 2018 Aug;63(8):1016-1023. doi: 10.4187/respcare.06031. Epub 2018 Jun 26. PMID 29945910
- [Background] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Roca O, Hernandez G, Diaz-Lobato S, Carratala JM, Gutierrez RM, Masclans JR; Spanish Multidisciplinary Group of High Flow Supportive Therapy in Adults (HiSpaFlow). Current evidence for the effectiveness of heated and humidified high flow nasal cannula supportive therapy in adult patients with respiratory failure. Crit Care. 2016 Apr 28;20(1):109. doi: 10.1186/s13054-016-1263-z. PMID 27121707
- See also: Drive Study link — https://drive.google.com/drive/u/0/folders/1D7-slVD5mPnbIMnCFT4j1JolktK9dBQ1